CLINICAL TRIAL: NCT00611026
Title: 12-Week, Randomized, Double-Blind, Double-Dummy, Placebo-Controlled, Parallel-Group, Multicenter Trial To Evaluate The Efficacy And Safety Of Fesoterodine In Comparison To Tolterodine ER In Patients With Overactive Bladder.
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of Fesoterodine in Comparison to Tolterodine Extended Release(ER)in Patients With Overactive Bladder.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A0221046
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Results first posted 2011-01-12 (Estimated); Last update posted 2011-02-02 (Estimated); Status verified 2011-01

CONDITIONS: Overactive Bladder
Keywords: Treatment of overactive bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Tolterodine Tartrate; fesoterodine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: Tolterodine ER
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo
- 3 (Experimental)
  Interventions: Drug: Fesoterodine

INTERVENTIONS:
Drug: Tolterodine ER — The tolterodine treatment will be 4 mg once daily(QD) for 12 weeks.
  Arms: 1
Drug: Placebo — Placebo treatment will be once daily(QD) for 12 weeks.
  Arms: 2
Drug: Fesoterodine — The fesoterodine treatment will start with 4 mg once daily(QD) for 1 week followed by a forced dose-escalation to 8mg once daily(QD) for 11 weeks.
  Arms: 3

SUMMARY:
To evaluate the efficacy and safety of fesoterodine in comparison to tolterodine and placebo for overactive bladder

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects with overactive bladder symptoms (subject-reported) for greater than or equal to 3 months prior to Screening/Enrollment visit.
* Reported at least an average of 1 UUI episode per 24 hours in the 3-day bladder diary prior to the Randomization/Baseline visit
* Mean urinary frequency of greater than or equal to 8 micturitions per 24 hours as verified by the 3-day bladder diary prior to randomization/Baseline visit.

Exclusion Criteria:

* Subjects with any condition that would contraindicate their usage of fesoterodine including: hypersensitivity to the active substance (fesoterodine fumarate) or to peanut or soya or any of the excipients, urinary retention, gastric retention, uncontrolled narrow angle glaucoma, myasthenia gravis, severe hepatic impairment (Child Pugh C), severe ulcerative colitis, and toxic megacolon.
* Subjects with clinically significant hepatic or renal disease or other significant unstable diseases.
* OAB symptoms caused by neurological conditions, known pathologies of urinary tract, etc.
* Subjects with previous history of acute urinary retention requiring catheterization, or severe voiding difficulties in the judgment of the investigator, prior to baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2417 (Actual)
Dates: Start 2008-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (194):
- United States (88):
  - Pfizer Investigational Site, Enterprise, Alabama
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Montgomery, Alabama
  - Pfizer Investigational Site, Chandler, Arizona
  - Pfizer Investigational Site, Peoria, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Clovis, California
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Upland, California
  - Pfizer Investigational Site, Vista, California
  - Pfizer Investigational Site, Westlake Village, California
  - Pfizer Investigational Site, Englewood, Colorado
  - Pfizer Investigational Site, New London, Connecticut
  - Pfizer Investigational Site, Bonita Spring, Florida
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Lake Worth, Florida
  - Pfizer Investigational Site, Leesburg, Florida
  - Pfizer Investigational Site, Longwood, Florida
  - Pfizer Investigational Site, Loxahatchee Groves, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Naples, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Stuart, Florida
  - Pfizer Investigational Site, Tallahassee, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Meridian, Idaho
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Peoria, Illinois
  - Pfizer Investigational Site, Avon, Indiana
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Noblesville, Indiana
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Bel Air, Maryland
  - Pfizer Investigational Site, North Dartmouth, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Royal Oak, Michigan
  - Pfizer Investigational Site, Troy, Michigan
  - Pfizer Investigational Site, Edina, Minnesota
  - Pfizer Investigational Site, Sartell, Minnesota
  - Pfizer Investigational Site, Olive Branch, Mississippi
  - Pfizer Investigational Site, Picayune, Mississippi
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Hamilton, New Jersey
  - Pfizer Investigational Site, Williamsville, New York
  - Pfizer Investigational Site, Cary, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Bensalem, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Uniontown, Pennsylvania
  - Pfizer Investigational Site, Cumberland, Rhode Island
  - Pfizer Investigational Site, Pawtucket, Rhode Island
  - Pfizer Investigational Site, Anderson, South Carolina
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Summerville, South Carolina
  - Pfizer Investigational Site, Johnson City, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, New Tazewell, Tennessee
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Bryan, Texas
  - Pfizer Investigational Site, Plano, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Sugar Land, Texas
  - Pfizer Investigational Site, Midvale, Utah
  - Pfizer Investigational Site, West Jordan, Utah
  - Pfizer Investigational Site, Arlington, Virginia
  - Pfizer Investigational Site, Charlottesville, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Virginia Beach, Virginia
  - Pfizer Investigational Site, Weber City, Virginia
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Spokane, Washington
- Brazil (6):
  - Pfizer Investigational Site, Salvador, Estado de Bahia
  - Pfizer Investigational Site, Goiânia, Goiás
  - Pfizer Investigational Site, Curitiba, Paraná
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo
- Bulgaria (5):
  - Pfizer Investigational Site, Pernik
  - Pfizer Investigational Site, Pleven
  - Pfizer Investigational Site, Plovdiv
  - Pfizer Investigational Site, Sofia
  - Pfizer Investigational Site, Veliko Tarnovo
- Canada (8):
  - Pfizer Investigational Site, Surrey, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Oshawa, Ontario
  - Pfizer Investigational Site, Chicoutimi, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Trois-Rivières, Quebec
  - Pfizer Investigational Site, Saskatoon, Saskatchewan
- Colombia (2):
  - Pfizer Investigational Site, Barranquilla, Atlántico
  - Pfizer Investigational Site, Bogotá, Colombia
- Costa Rica (3):
  - Pfizer Investigational Site, Alajuela, Alajuela Province
  - Pfizer Investigational Site, Cartago, Cartago Province
  - Pfizer Investigational Site, San José, Provincia de San José
- Estonia (2):
  - Pfizer Investigational Site, Tallinn
  - Pfizer Investigational Site, Tartu
- Germany (8):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Grünstadt
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Krumbach
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Marburg
  - Pfizer Investigational Site, Muelheim A.d. Ruhr
  - Pfizer Investigational Site, München
- Greece (5):
  - Pfizer Investigational Site, Heraklion/Voutes, Crete
  - Pfizer Investigational Site, Alexandroupoli
  - Pfizer Investigational Site, Athens, Maroussi
  - Pfizer Investigational Site, Larissa
  - Pfizer Investigational Site, Thessaloniki
- Hungary (5):
  - Pfizer Investigational Site, Debrecen
  - Pfizer Investigational Site, Győr
  - Pfizer Investigational Site, Nyíregyháza
  - Pfizer Investigational Site, Salgótarján
  - Pfizer Investigational Site, Szentes
- India (6):
  - Pfizer Investigational Site, Hyderabad, Andhra Pradesh
  - Pfizer Investigational Site, Ahmedabad, Gujarat
  - Pfizer Investigational Site, Nadiād, Gujarat
  - Pfizer Investigational Site, Bengaluru, Karnataka
  - Pfizer Investigational Site, Pune, Maharashtra
  - Pfizer Investigational Site, New Delhi
- Ireland (2):
  - Pfizer Investigational Site, Beaumont, Dublin
  - Pfizer Investigational Site, Dublin
- Pfizer Investigational Site, Riga, Latvia
- Lithuania (3):
  - Pfizer Investigational Site, Kaunas
  - Pfizer Investigational Site, Klaipėda
  - Pfizer Investigational Site, Vilnius
- Pfizer Investigational Site, Kuala Lumpur, Malaysia
- Poland (7):
  - Pfizer Investigational Site, Bialystok
  - Pfizer Investigational Site, Bydgoszcz
  - Pfizer Investigational Site, Gdynia
  - Pfizer Investigational Site, Krakow
  - Pfizer Investigational Site, Lublin
  - Pfizer Investigational Site, Poznan
  - Pfizer Investigational Site, Słupsk
- Romania (4):
  - Pfizer Investigational Site, Bucharest, București
  - Pfizer Investigational Site, Bucharest, Sector 5,
  - Pfizer Investigational Site, Sibiu, Sibiu County
  - Pfizer Investigational Site, Arad
- Russia (3):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Rostov-on-Don
  - Pfizer Investigational Site, Saint Petersburg
- Pfizer Investigational Site, Singapore, Singapore, Singapore
- Slovakia (5):
  - Pfizer Investigational Site, Nitra
  - Pfizer Investigational Site, Považská Bystrica
  - Pfizer Investigational Site, Prešov
  - Pfizer Investigational Site, Trenčín
  - Pfizer Investigational Site, Zvolen
- South Africa (7):
  - Pfizer Investigational Site, Claremont, Cape Town
  - Pfizer Investigational Site, Bloemfontein, Free State
  - Pfizer Investigational Site, Vosloorus, Gauteng
  - Pfizer Investigational Site, Durban, KwaZulu-Natal
  - Pfizer Investigational Site, Pietermaritzburg, KwaZulu-Natal
  - Pfizer Investigational Site, Pretoria
  - Pfizer Investigational Site, Roodepoort
- South Korea (6):
  - Pfizer Investigational Site, Jeonju, Jeollabuk-do
  - Pfizer Investigational Site, Busan
  - Pfizer Investigational Site, Daegu
  - Pfizer Investigational Site, Incheon
  - Pfizer Investigational Site, Seoul
  - Pfizer Investigational Site, Suwon
- Spain (5):
  - Pfizer Investigational Site, Santander, Cantabria
  - Pfizer Investigational Site, Las Palmas de Gran Canaria, Las Palmas de Gran Canaria
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, San Cristóbal de La Laguna, Santa Cruz de Tenerife
  - Pfizer Investigational Site, Valencia, Valencia
- Sweden (6):
  - Pfizer Investigational Site, Karlskoga
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Norrköping
  - Pfizer Investigational Site, Örebro
  - Pfizer Investigational Site, Skövde
  - Pfizer Investigational Site, Stockholm
- Ukraine (5):
  - Pfizer Investigational Site, Chernivtsi
  - Pfizer Investigational Site, Dnipropetrovsk
  - Pfizer Investigational Site, Kyiv
  - Pfizer Investigational Site, Uzhhorod
  - Pfizer Investigational Site, Zaporizhzhia

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- [Derived] Wagg AS, Herschorn S, Carlsson M, Fernet M, Oelke M. A plain language summary of the likelihood of symptom relief for patients taking fesoterodine for overactive bladder. J Comp Eff Res. 2022 Sep;11(13):919-925. doi: 10.2217/cer-2022-0041. Epub 2022 Jul 26. PMID 35881009
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221046&StudyName=Clinical%20Trial%20to%20Evaluate%20the%20Efficacy%20and%20Safety%20of%20Fesoterodine%20in%20Comparison%20to%20Tolterodine%20ER%20in%20Patients%20with%20Overactive%20Bladder.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with urgency incontinence Overactive Bladder (OAB) symptoms who met all entrance criteria were randomized to the double-blind treatment period.
Pre-assignment Details: 3867 participants entered the single-blind placebo run-in period; 2417 participants completed single-blind placebo run-in and progressed to randomization in the double-blind treatment period.
Groups:
- Placebo: Tablets 4 milligrams (mg) orally (PO) once daily (QD) for 1 week followed by a forced dose escalation to 8 mg PO QD for 11 weeks or capsules (4 mg) PO QD for 12 weeks matching to treatment.
- Tolterodine ER: Capsules 4 mg PO QD for 12 weeks. Tolterodine Extended Release (ER).
- Fesoterodine: Tablets 4 mg PO QD for 1 week followed by a forced dose escalation to 8 mg PO QD for 11 weeks.
Period: Randomized to Double-blind Treatment
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Started | 480 | 974 | 963
Completed | 478 | 973 | 960
Not Completed | 2 | 1 | 3
Not completed — Not treated | 2 | 1 | 3
Period: Double-blind Treatment Period
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Started | 478 | 973 | 960
Completed | 431 | 885 | 862
Not Completed | 47 | 88 | 98
Not completed — Death | 1 | 0 | 0
Not completed — Adverse Event | 9 | 28 | 46
Not completed — Lack of Efficacy | 11 | 10 | 4
Not completed — Lost to Follow-up | 6 | 11 | 14
Not completed — Withdrawal by Subject | 7 | 19 | 16
Not completed — Other | 13 | 20 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tolterodine ER | Fesoterodine | Total
Number analyzed (Participants) | 478 | 973 | 960 | 2411
Age, Customized [Number; unit: participants]
  Between 18 and 44 years | 70 | 157 | 156 | 383
  Between 45 and 64 years | 214 | 462 | 474 | 1150
  ≥65 years | 194 | 354 | 330 | 878
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 410 | 818 | 816 | 2044
  Male | 68 | 155 | 144 | 367

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Number of Urgency Urinary Incontinence (UUI) Episodes Per 24 Hours at Week 12
Description: UUI per 24 hours: total number of micturitions with Urinary Sensation Scale (USS) of 5 divided by total number of diary days collected at visit. USS: 5-item scale to measure urinary urgency; range: 1 (no feeling of urgency) to 5 (unable to hold; leak urine).
Time Frame: Baseline, Week 12
Population: Full analysis set (FAS): at least 1 dose of assigned treatment, data for at least 1 baseline or post-baseline efficacy assessment, and excluded 77 participants from 3 study sites with Good Clinical Practices (GCP) deviations (Fesoterodine N=30, Tolterodine ER N=31, Placebo N=16). Decision to exclude that data was made while the study was blinded.
Measure: Mean (Standard Error); unit: episodes per 24 hours
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 448 | 926 | 908
episodes per 24 hours | -1.62 (0.07) | -1.74 (0.06) | -1.95 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine versus (vs) placebo at Week 12. Treatment effects estimated by Winsorized means (5% of the tails were censored, ie, replaced with the value at the fifth (5th) and ninety-fifth (95th) percentile, respectively). If normality assumptions were severely violated (proportion of non normal observations > 5%) a non-parametric analysis was to be conducted using Van Elteren's test stratified by baseline quartile of the diary variable analyzed; Test type: Superiority or Other; p < 0.0001, Van Elteren's Test — Comparison fesoterodine vs tolterodine ER performed only if statistical significance favoring fesoterodine achieved for fesoterodine vs placebo to preserve overall alpha level at 5%; pairwise comparison also performed for tolterodine ER vs placebo; P-value based on Van Elteren's Test (a stratified Wilcoxon-Mann Whitney test) adjusted by baseline UUI quartile
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment difference tolterodine ER vs placebo at Week 12. Treatment effects estimated by Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95th percentile, respectively); Test type: Superiority or Other; p = 0.0228, Van Elteren's Test — [p-value comment as in outcome 1, analysis 1]; P-value based on Van Elteren's Test (a stratified Wilcoxon-Mann Whitney test) adjusted by baseline UUI quartile
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference fesoterodine vs tolterodine ER at Week 12. Treatment effects estimated by Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95th percentile, respectively); Test type: Superiority or Other; p = 0.0072, Van Elteren's test — [p-value comment as in outcome 1, analysis 1]; P-value based on Van Elteren's Test (a stratified Wilcoxon-Mann Whitney test) adjusted by baseline UUI quartile

2. Secondary Outcome: Change From Baseline in Mean Voided Volume Per Micturition
Description: Mean voided volume in milliliters (mL) calculated as sum of voided volume divided by the total number of micturition episodes with a recorded voided volume greater than 0 in the 3-day diary at that visit.
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: FAS; (n)=number of participants with non-missing numerical change from baseline to the respective post-baseline value (Week 1, Week 4 [Last Observation Carried Forward (LOCF)], or Week 12 [LOCF]) for placebo, tolterodine ER, and fesoterodine, respectively.
Measure: Mean (Standard Error); unit: mL
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 452 | 930 | 912
mL
  Week 1 (n=447, 917, 895) | 9.80 (1.92) | 15.65 (1.43) | 18.63 (1.55)
  Week 4 [LOCF] (n=452, 927, 909) | 14.27 (2.28) | 26.43 (1.76) | 32.26 (1.94)
  Week 12 [LOCF] (n=452, 930, 912) | 17.34 (2.40) | 28.43 (1.82) | 34.47 (2.06)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 1. Treatment effects estimated by Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95th percentile, respectively). If normality assumptions were severely violated (proportion of non normal observations > 5%) a non-parametric analysis was to be conducted using Van Elteren's test stratified by baseline quartile of the diary variable analyzed; Test type: Superiority or Other; p = 0.0020, Van Elteren's Test; P-value based on Van Elteren's Test (a stratified Wilcoxon-Mann Whitney test) adjusted by baseline quartile of voided volume
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment difference tolterodine ER vs placebo at Week 1. Treatment effects estimated by Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95th percentile, respectively); Test type: Superiority or Other; p = 0.0519, Van Elteren's Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference fesoterodine vs tolterodine ER at Week 1. Treatment effects estimated by Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95th percentile, respectively); Test type: Superiority or Other; p = 0.1503, Van Elteren's Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 4. Treatment effects estimated by Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95th percentile, respectively); Test type: Superiority or Other; p < 0.0001, Van Elteren's Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Tolterodine ER; Treatment difference tolterodine ER vs placebo at Week 4. Treatment effects estimated by Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95th percentile, respectively); Test type: Superiority or Other; p = 0.0002, Van Elteren's Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference fesoterodine vs tolterodine ER at Week 4. Treatment effects estimated by Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95th percentile, respectively); Test type: Superiority or Other; p = 0.0130, Van Elteren's; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 12. Treatment effects estimated by Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95th percentile, respectively); Test type: Superiority or Other; p < 0.0001, Van Elteren's Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs Tolterodine ER; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0021, Van Elteren's Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: Tolterodine ER vs Fesoterodine; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.0525, Van Elteren's Test; [statistical method as in outcome 2, analysis 1]

3. Secondary Outcome: Change From Baseline in Mean Number of Micturitions Per 24 Hours
Description: The mean number of micturitions was calculated as the total number of micturitions divided by the total number of diary days collected at that visit.
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: FAS; (n)=number of participants with non-missing numerical change from baseline to the respective post-baseline value (Week 1, Week 4 [LOCF], or Week 12 [LOCF]) for placebo, tolterodine ER, and fesoterodine, respectively.
Measure: Least Squares Mean (Standard Error); unit: micturitions per 24 hours
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 454 | 935 | 916
micturitions per 24 hours
  Week 1 (n=448, 921, 908) | -0.8 (0.1) | -1.0 (0.1) | -1.0 (0.1)
  Week 4 [LOCF] (n=454, 931, 916) | -1.5 (0.1) | -1.8 (0.1) | -2.1 (0.1)
  Week 12 [LOCF] (n=454, 935, 916) | -2.0 (0.1) | -2.3 (0.1) | -2.6 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 1; Test type: Superiority or Other; p = 0.0161, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.5 to -0.1], Standard Error of Mean 0.1 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 1; Test type: Superiority or Other; p = 0.0944, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to 0.0], Standard Error of Mean 0.1 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference fesoterodine vs Tolterodine ER at Week 1; Test type: Superiority or Other; p = 0.3613, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.3 to 0.1], Standard Error of Mean 0.1 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-0.9 to -0.4], Standard Error of Mean 0.1 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 5: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 4; Test type: Superiority or Other; p = 0.0043, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.6 to -0.1], Standard Error of Mean 0.1 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 6: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference fesoterodine vs Tolterodine ER at Week 4; Test type: Superiority or Other; p = 0.0186, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.5 to -0.0], Standard Error of Mean 0.1 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 7: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-0.9 to -0.4], Standard Error of Mean 0.1 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 8: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 12; Test type: Superiority or Other; p = 0.0407, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.6 to -0.0], Standard Error of Mean 0.1 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 9: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference fesoterodine vs Tolterodine ER at Week 12; Test type: Superiority or Other; p = 0.0016, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.6 to -0.1], Standard Error of Mean 0.1 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean

4. Secondary Outcome: Percent Change From Baseline of Micturitions Per 24 Hours
Description: Percent change of micturitions per 24 hours was calculated as change in 24-hour mean at that visit divided by the baseline 24-hour mean multiplied by 100 (ie, 100%*(Week 1 or 4 or 12 - baseline)/baseline).
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: FAS; (n)=number of participants with non-missing percent change from baseline to the respective post-baseline value (Week 1, Week 4 [LOCF], or Week 12 [LOCF]) for placebo, tolterodine ER, and fesoterodine, respectively.
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 454 | 935 | 916
percent change
  Week 1 (n=448, 921, 908) | -7.1 [-70.6 to 53.6] | -9.4 [-64.3 to 74.2] | -9.0 [-61.9 to 89.3]
  Week 4 [LOCF] (n=454, 931, 916) | -13.4 [-64.4 to 118.8] | -16.7 [-67.9 to 64.0] | -18.9 [-68.8 to 96.2]
  Week 12 [LOCF] (n=454, 935, 916) | -18.2 [-66.7 to 118.8] | -20.8 [-67.5 to 70.8] | -23.5 [-75.3 to 64.3]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 1; Test type: Superiority or Other; p = 0.0217, ANCOVA — Inferential testing: percent change from baseline only carried out for given end/time point if corresponding numeric change result statistically significant (to preserve alpha level at 5% within each type of diary endpoint for a given comparison); Based on a ranked analysis of covariance model with country and treatment as factors, and ranked baseline value as a covariate
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 4; Test type: Superiority or Other; p = 0.0020, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference fesoterodine vs Tolterodine ER at Week 4; Test type: Superiority or Other; p = 0.0217, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 12; Test type: Superiority or Other; p = 0.0421, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference fesoterodine vs Tolterodine ER at Week 12; Test type: Superiority or Other; p = 0.0023, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 4, analysis 1]

5. Secondary Outcome: Change From Baseline in Mean Number of Nocturnal Micturitions Per 24 Hours
Description: Mean number of nocturnal micturitions per 24 hours was calculated as the total number of all micturitions divided by the total number of diary days collected at that visit. Nocturnal micturitions are those recorded in the Bedtime section of the diary. Nocturnal (Bedtime) was defined as the time the participant went to bed until he/she arose to start the next day.
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: FAS; (n)=number of participants with baseline nocturnal micturitions >0 per 24 hours and non-missing change from baseline to the respective post-baseline value (Week 1, Week 4 [LOCF], or Week 12 [LOCF]) for placebo, tolterodine ER, and fesoterodine, respectively.
Measure: Least Squares Mean (Standard Error); unit: nocturnal micturitions per 24 hours
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 445 | 899 | 892
nocturnal micturitions per 24 hours
  Week 1 (n=432, 879, 871) | -0.2 (0.1) | -0.3 (0.0) | -0.3 (0.0)
  Week 4 [LOCF] (n=437, 888, 879) | -0.4 (0.1) | -0.5 (0.0) | -0.5 (0.0)
  Week 12 [LOCF] (n=437, 892, 879) | -0.5 (0.1) | -0.6 (0.0) | -0.7 (0.0)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 1; Test type: Superiority or Other; p = 0.3823, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.1 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 1; Test type: Superiority or Other; p = 0.4802, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.1 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference fesoterodine vs Tolterodine ER at Week 1; Test type: Superiority or Other; p = 0.8355, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.0 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 4; Test type: Superiority or Other; p = 0.0286, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.12 to -0.0], Standard Error of Mean 0.1 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 5: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 4; Test type: Superiority or Other; p = 0.0794, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.2 to 0.0], Standard Error of Mean 0.1 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 6: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference fesoterodine vs Tolterodine ER at Week 4; Test type: Superiority or Other; p = 0.5906, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.0 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 7: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p = 0.0134, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.3 to -0.0], Standard Error of Mean 0.1 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 8: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 12; Test type: Superiority or Other; p = 0.1759, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.2 to 0.0], Standard Error of Mean 0.1 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 9: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference fesoterodine vs Tolterodine ER at Week 12; Test type: Superiority or Other; p = 0.1661, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.2 to 0.0], Standard Error of Mean 0.0 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean

6. Secondary Outcome: Percent Change From Baseline of Nocturnal Micturitions Per 24 Hours
Description: Percent change of nocturnal micturitions per 24 hours was calculated as change in 24-hour mean at that visit divided by the baseline 24-hour mean multiplied by 100 (ie, 100%*(Week 1 or 4 or 12 - baseline)/baseline). Nocturnal micturitions are those recorded in the Bedtime section of the diary. Nocturnal (Bedtime) was defined as the time the participant went to bed until he/she arose to start the next day.
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: as for outcome 5
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 445 | 899 | 892
percent change
  Week 1 (n=432, 879, 871) | -7.7 [-100.0 to 500.0] | -14.3 [-100.0 to 500.0] | -12.5 [-100.0 to 800.0]
  Week 4 [LOCF] (n=437, 888, 879) | -20.0 [-100.0 to 600.0] | -25.0 [-100.0 to 400.0] | -25.0 [-100.0 to 1600.0]
  Week 12 [LOCF] (n=437, 892, 879) | -27.3 [-100.0 to 800.0] | -33.3 [-100.0 to 350.0] | -33.3 [-100.0 to 500.0]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 4; Test type: Superiority or Other; p = 0.0021, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Based on a ranked analysis of covariance model with terms for country and treatment and ranked baseline value as a covariate
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p = 0.0200, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 6, analysis 1]

7. Secondary Outcome: Change From Baseline in Mean Number of Urgency Urinary Incontinence (UUI) Episodes Per 24 Hours at Week 1 and Week 4
Description: UUI episodes per 24 hours calculated as total number of micturitions with Urinary Sensation Scale (USS) of 5 divided by total number of diary days collected at visit. USS is 5-item scale measuring urinary urgency; range is 1 (no feeling of urgency) to 5 (unable to hold; leak urine).
Time Frame: Baseline, Week 1, Week 4
Population: FAS; (n)=number of participants with baseline UUI >0 per 24 hours and non-missing change from baseline to respective post-baseline value (Week 1 or Week 4 [LOCF] for placebo, tolterodine ER, and fesoterodine, respectively.
Measure: Mean (Standard Error); unit: episodes per 24 hours
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 456 | 932 | 920
episodes per 24 hours
  Week 1 (n=442, 911, 899) | -0.80 (0.06) | -0.95 (0.05) | -1.03 (0.05)
  Week 4 [LOCF] (n=448, 922, 908) | -1.31 (0.07) | -1.52 (0.05) | -1.68 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 1. Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95th percentile, respectively). If normality assumptions were severely violated (proportion of non normal observations > 5%) a non-parametric analysis was to be conducted using Van Elteren's test stratified by baseline quartile of the diary variable analyzed; Test type: Superiority or Other; p = 0.0006, Van Elteren's Test; P-value based on Van Elteren's Test (a stratified Wilcoxon-Mann Whitney test) adjusted by baseline UUI quartile
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 1. Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95th percentile, respectively); Test type: Superiority or Other; p = 0.0202, Van Elteren's Test; P-value based on Van Elteren's Test (a stratified Wilcoxon-Mann Whitney test) adjusted by baseline UUI quartile
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference fesoterodine vs Tolterodine ER at Week 1. Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95th percentile, respectively); Test type: Superiority or Other; p = 0.2126, Van Elteren's Test; P-value based on Van Elteren's Test (a stratified Wilcoxon-Mann Whitney test) adjusted by baseline UUI quartile
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 4. Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95th percentile, respectively); Test type: Superiority or Other; p < 0.0001, Van Elteren's Test; P-value based on Van Elteren's Test (a stratified Wilcoxon-Mann Whitney test) adjusted by baseline UUI quartile
Statistical Analysis 5: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 4. Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95th percentile, respectively); Test type: Superiority or Other; p = 0.0019, Van Elteren's Test; P-value based on Van Elteren's Test (a stratified Wilcoxon-Mann Whitney test) adjusted by baseline UUI quartile
Statistical Analysis 6: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference fesoterodine vs Tolterodine ER at Week 4. Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95th percentile, respectively); Test type: Superiority or Other; p = 0.0148, Van Elteren's Test; P-value based on Van Elteren's Test (a stratified Wilcoxon-Mann Whitney test) adjusted by baseline UUI quartile

8. Secondary Outcome: Percent Change From Baseline of UUI Episodes Per 24 Hours
Description: UUI episodes per 24 hours calculated as total number of micturitions with USS of 5 in diary. USS is 5-item scale measuring urinary urgency; range is
  1 (no feeling of urgency) to 5 (unable to hold; leak urine). Change calculated as UUI episodes per 24 hours at observation divided by baseline number of UUI episodes per 24 hours, multiplied by 100.
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: FAS; (n)=number of participants with baseline UUI >0 per 24 hours and non-missing change from baseline to respective post-baseline value (Week 1, Week 4 [LOCF], or Week 12 [LOCF]) for placebo, tolterodine ER, and fesoterodine, respectively.
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 456 | 932 | 920
percent change
  Week 1 (n=442, 911, 899) | -40.8 [-100.0 to 966.7] | -50.0 [-100.0 to 366.7] | -50.0 [-100.0 to 633.3]
  Week 4 [LOCF] (n=448, 922, 908) | -75.0 [-100.0 to 1000.0] | -88.9 [-100.0 to 900.0] | -100.0 [-100.0 to 666.7]
  Week 12 [LOCF] (n=448, 926, 908) | -100.0 [-100.0 to 612.5] | -100.0 [-100.0 to 687.5] | -100.0 [-100.0 to 500.0]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 1; Test type: Superiority or Other; p = 0.0012, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 1; Test type: Superiority or Other; p = 0.0205, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 4; Test type: Superiority or Other; p = 0.0038, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference Tolterodine ER vs Fesoterodine at Week 4; Test type: Superiority or Other; p = 0.0219, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p = 0.0001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 12; Test type: Superiority or Other; p = 0.0805, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 8: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference Tolterodine ER vs Fesoterodine at Week 12; Test type: Superiority or Other; p = 0.0093, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 6, analysis 1]

9. Secondary Outcome: Change From Baseline in Mean Number of Urgency Urinary Episodes Per 24 Hours (Urinary Sensation Scale ≥3 in the Diary)
Description: Urgency Urinary episodes per 24 hours: total number of micturitions with Urinary Sensation Scale (USS) of ≥3 divided by total number of diary days collected at visit. USS: 5-item scale to measure urinary urgency; range: 1 (no feeling of urgency) to 5 (unable to hold; leak urine).
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: FAS; (n)=number of participants with baseline urgency episodes >0 per 24 hours and non-missing numerical change from baseline to the respective post-baseline value (Week 1, Week 4 [LOCF], or Week 12 [LOCF]) for placebo, tolterodine ER, and fesoterodine, respectively.
Measure: Least Squares Mean (Standard Error); unit: episodes per 24 hours
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 461 | 940 | 928
episodes per 24 hours
  Week 1 (n=447, 918, 906) | -0.8 (0.2) | -1.0 (0.1) | -1.2 (0.2)
  Week 4 [LOCF] (n=453, 929, 915) | -1.9 (0.2) | -2.5 (0.2) | -3.1 (0.2)
  Week 12 [LOCF] (n=453, 933, 915) | -3.2 (0.2) | -3.5 (0.2) | -4.2 (0.2)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 1; Test type: Superiority or Other; p = 0.0374, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.7 to -0.0], Standard Error of Mean 0.2 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 1; Test type: Superiority or Other; p = 0.3161, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.2], Standard Error of Mean 0.2 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference Tolterodine ER vs Fesoterodine at Week 1; Test type: Superiority or Other; p = 0.1817, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.1], Standard Error of Mean 0.1 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-1.6 to -0.8], Standard Error of Mean 0.2 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 5: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 4; Test type: Superiority or Other; p = 0.0054, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.0 to -0.2], Standard Error of Mean 0.2 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 6: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference Tolterodine ER vs Fesoterodine at Week 4; Test type: Superiority or Other; p = 0.0005, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-0.9 to -0.3], Standard Error of Mean 0.2 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 7: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-1.5 to -0.6], Standard Error of Mean 0.2 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 8: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 12; Test type: Superiority or Other; p = 0.1467, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.7 to 0.1], Standard Error of Mean 0.2 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 9: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference Tolterodine ER vs Fesoterodine at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.1 to -0.4], Standard Error of Mean 0.2 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean

10. Secondary Outcome: Percent Change From Baseline in Mean Number of Urgency Urinary Episodes Per 24 Hours (Urinary Sensation Scale ≥3 in the Diary)
Description: Percent change from baseline in mean number of Urgency Urinary episodes per 24 hours (Urinary Sensation Scale ≥3 in the diary). Change calculated as UUI episodes per 24 hours at observation divided by baseline number of UUI episodes per 24 hours, multiplied by 100.
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: as for outcome 9
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 461 | 940 | 928
percent change
  Week 1 (n=447, 918, 906) | -9.4 [-100.0 to 385.7] | -12.0 [-100.0 to 325.0] | -11.8 [-100.0 to 433.3]
  Week 4 [LOCF] (n=453, 929, 915) | -17.2 [-100.0 to 457.1] | -26.3 [-100.0 to 350.0] | -32.1 [-100.0 to 433.3]
  Week 12 [LOCF] (n=453, 933, 915) | -31.0 [-100.0 to 385.7] | -37.5 [-100.0 to 475.0] | -45.5 [-100.0 to 266.7]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 1; Test type: Superiority or Other; p = 0.0828, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 4; Test type: Superiority or Other; p = 0.0008, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference Tolterodine ER vs Fesoterodine at Week 4; Test type: Superiority or Other; p = 0.0022, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference Tolterodine ER vs Fesoterodine at Week 12; Test type: Superiority or Other; p = 0.0008, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 6, analysis 1]

11. Secondary Outcome: Change From Baseline in Mean Number of Severe Urgency Episodes Per 24 Hours
Description: Mean number of severe urgency episodes (USS rating ≥4 in diary ) per 24 hours calculated as the total number of micturitions with USS ≥4 divided by total number of diary days collected at that visit. USS: 5-item scale to measure urinary urgency; range: 1 (no feeling of urgency) to 5 (unable to hold; leak urine).
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: FAS; (n)=number of participants with baseline severe urgency episodes >0 per 24 hours and non-missing change from baseline to the respective post-baseline value (Week 1, Week 4 [LOCF], or Week 12 [LOCF]) for placebo, tolterodine ER, and fesoterodine, respectively.
Measure: Mean (Standard Error); unit: severe urgency episodes per 24 hours
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 460 | 937 | 924
severe urgency episodes per 24 hours
  Week 1 (n=446, 915, 902) | -1.14 (0.13) | -1.34 (0.10) | -1.58 (0.11)
  Week 4 [LOCF] (n=452, 926, 911) | -2.14 (0.16) | -2.71 (0.12) | -3.21 (0.12)
  Week 12 [LOCF] (n=452, 930, 911) | -3.01 (0.17) | -3.39 (0.13) | -4.08 (0.13)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 1. Treatment effects estimated by Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95 percentile, respectively). If normality assumptions were severely violated (proportion of non normal observations > 5%) a non-parametric analysis was to be conducted using Van Elteren's test stratified by baseline quartile of the diary variable analyzed; Test type: Superiority or Other; p = 0.0576, Van Elteren's Test; P-value based on Van Elteren's Test (a stratified Wilcoxon-Mann Whitney test) adjusted by baseline quartile of severe urgency episodes
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 1. Treatment effects estimated by Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95 percentile, respectively); Test type: Superiority or Other; p = 0.2230, Van Elteren's Test; [statistical method as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference fesoterodine vs Tolterodine ER at Week 1. Treatment effects estimated by Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95 percentile, respectively); Test type: Superiority or Other; p = 0.3555, Van Elteren's Test; [statistical method as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 4. Treatment effects estimated by Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95 percentile, respectively); Test type: Superiority or Other; p < 0.0001, Van Elteren's Test; [statistical method as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 4. Treatment effects estimated by Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95 percentile, respectively); Test type: Superiority or Other; p = 0.0009, Van Elteren's Test; [statistical method as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference fesoterodine vs Tolterodine ER at Week 4. Treatment effects estimated by Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95 percentile, respectively); Test type: Superiority or Other; p = 0.0071, Van Elteren's Test; [statistical method as in outcome 11, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 12. Treatment effects estimated by Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95 percentile, respectively); Test type: Superiority or Other; p < 0.0001, Van Elteren's Test; [statistical method as in outcome 11, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 12. Treatment effects estimated by Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95 percentile, respectively); Test type: Superiority or Other; p = 0.1764, Van Elteren's Test; [statistical method as in outcome 11, analysis 1]
Statistical Analysis 9: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference fesoterodine vs Tolterodine ER at Week 12. Treatment effects estimated by Winsorized means (5% of the tails were censored, ie, replaced with the value at the 5th and 95 percentile, respectively); Test type: Superiority or Other; p = 0.0001, Van Elteren's Test; [statistical method as in outcome 11, analysis 1]

12. Secondary Outcome: Percent Change From Baseline of Severe Urgency Episodes Per 24 Hours
Description: Percent change calculated as change in severe urgency episodes (USS rating ≥4 in diary ) per 24 hours at that visit divided by the baseline number of severe urgency episodes per 24 hours, multiplied by 100. USS is 5-item scale measuring urinary urgency; range is 1 (no feeling of urgency) to 5 (unable to hold; leak urine).
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: as for outcome 11
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 460 | 937 | 924
percent change
  Week 1 (n=446, 915, 902) | -19.7 [-100.0 to 575.0] | -24.1 [-100.0 to 500.0] | -25.0 [-100.0 to 475.0]
  Week 4 [LOCF] (n=452, 926, 911) | -41.7 [-100.0 to 533.3] | -55.6 [-100.0 to 800.0] | -61.1 [-100.0 to 433.3]
  Week 12 [LOCF] (n=452, 930, 911) | -61.0 [-100.0 to 1850.0] | -69.2 [-100.0 to 600.0] | -79.3 [-100.0 to 440.0]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 4; Test type: Superiority or Other; p = 0.0003, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference Tolterodine ER vs Fesoterodine at Week 4; Test type: Superiority or Other; p = 0.0302, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference Tolterodine ER vs Fesoterodine at Week 12; Test type: Superiority or Other; p = 0.0007, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 6, analysis 1]

13. Secondary Outcome: Change From Baseline in Mean Urinary Sensation Scale (USS) Rating Per Micturition Per 24 Hours.
Description: Mean USS rating calculated as the sum of rating scores on USS per 24 hours divided by the total number of micturitions per 24 hours with non-missing rating at that visit. USS is 5-item scale measuring urinary urgency; range is 1 (no feeling of urgency) to 5 (unable to hold; leak urine).
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 453 | 933 | 915
scores on a scale
  Week 1 (n=447, 918, 906) | -0.2 (0.0) | -0.2 (0.0) | -0.2 (0.0)
  Week 4 [LOCF] (n=453, 929, 915) | -0.3 (0.0) | -0.4 (0.0) | -0.5 (0.0)
  Week 12 [LOCF] (n=453, 933, 915) | -0.6 (0.0) | -0.6 (0.0) | -0.7 (0.0)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 1; Test type: Superiority or Other; p = 0.0701, ANCOVA; Based on an analysis of covariance model with terms for country and treatment with baseline value as a covariate; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.1 to 0.0], Standard Error of Mean 0.0 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 1; Test type: Superiority or Other; p = 0.4823, ANCOVA; Based on an analysis of covariance model with terms for country and treatment with baseline value as a covariate; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.1 to 0.0], Standard Error of Mean 0.0 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference Tolterodine ER vs Fesoterodine at Week 1; Test type: Superiority or Other; p = 0.1702, ANCOVA; Based on an analysis of covariance model with terms for country and treatment with baseline value as a covariate; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.1 to 0.0], Standard Error of Mean 0.0 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA; Based on an analysis of covariance model with terms for country and treatment with baseline value as a covariate; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.3 to -0.1], Standard Error of Mean 0.0 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 5: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 4; Test type: Superiority or Other; p = 0.0059, ANCOVA; Based on an analysis of covariance model with terms for country and treatment with baseline value as a covariate; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to -0.0], Standard Error of Mean 0.0 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 6: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference Tolterodine ER vs Fesoterodine at Week 4; Test type: Superiority or Other; p = 0.0014, ANCOVA; Based on an analysis of covariance model with terms for country and treatment with baseline value as a covariate; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to -0.0], Standard Error of Mean 0.0 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 7: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; Based on an analysis of covariance model with terms for country and treatment with baseline value as a covariate; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.3 to -0.1], Standard Error of Mean 0.0 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 8: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 12; Test type: Superiority or Other; p = 0.3110, ANCOVA; Based on an analysis of covariance model with terms for country and treatment with baseline value as a covariate; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.1 to 0.0], Standard Error of Mean 0.0 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 9: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference Tolterodine ER vs Fesoterodine at Week 12; Test type: Superiority or Other; p = 0.0004, ANCOVA; Based on an analysis of covariance model with terms for country and treatment with baseline value as a covariate; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to -0.1], Standard Error of Mean 0.0 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean

14. Secondary Outcome: Change From Baseline in Frequency-Urgency Sum (FUS) Per 24 Hours (Synonymous With USS Sum in the Study Protocol)
Description: Frequency-Urgency Sum per 24 hours calculated as mean rating scores on the USS multiplied by the mean number of micturitions per 24 hours at that visit. USS is 5-item scale measuring urinary urgency; range is 1 (no feeling of urgency) to 5 (unable to hold; leak urine).
Time Frame: Baseline, Week 1, Week 4, Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 453 | 933 | 915
scores on a scale
  Week 1 (n=447, 918, 906) | -4.0 (0.6) | -4.8 (0.5) | -5.5 (0.5)
  Week 4 [LOCF] (n=453, 929, 915) | -8.1 (0.7) | -10.1 (0.6) | -12.0 (0.6)
  Week 12 [LOCF] (n=453, 933, 915) | -12.0 (0.7) | -13.2 (0.6) | -15.6 (0.6)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 1; Test type: Superiority or Other; p = 0.0136, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and baseline value as a covariate; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-2.7 to -0.3], Standard Error of Mean 0.6 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 1; Test type: Superiority or Other; p = 0.1918, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and baseline value as a covariate; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-2.0 to 0.4], Standard Error of Mean 0.6 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference Tolterodine ER vs Fesoterodine at Week 1; Test type: Superiority or Other; p = 0.1505, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and baseline value as a covariate; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.7 to 0.3], Standard Error of Mean 0.5 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and baseline value as a covariate; Mean Difference (Final Values) = -3.9, 95% CI 2-sided [-5.2 to -2.6], Standard Error of Mean 0.7 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 5: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 4; Test type: Superiority or Other; p = 0.0034, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and baseline value as a covariate; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-3.3 to -0.7], Standard Error of Mean 0.7 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 6: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference Tolterodine ER vs Fesoterodine at Week 4; Test type: Superiority or Other; p = 0.0006, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and baseline value as a covariate; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-3.0 to -0.8], Standard Error of Mean 0.5 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 7: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and baseline value as a covariate; Mean Difference (Final Values) = -3.7, 95% CI 2-sided [-5.0 to -2.3], Standard Error of Mean 0.7 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 8: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 12; Test type: Superiority or Other; p = 0.0859, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and baseline value as a covariate; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.5 to 0.2], Standard Error of Mean 0.7 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 9: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference Tolterodine ER vs Fesoterodine at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and baseline value as a covariate; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-3.6 to -1.4], Standard Error of Mean 0.6 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean

15. Secondary Outcome: Diary Dry Rate: Percentage of Participants With no Urgency Urinary Incontinence (UUI) in the 3-day Bladder Diary
Description: Diary dry rate: percentage of participants with no urgency urinary incontinence episode reported in the 3 day diary at the respective time-point; based on USS: 5-item scale measuring urinary urgency; range is 1 (no feeling of urgency) to 5 (unable to hold; leak urine).
Time Frame: Week 1, Week 4, Week 12
Population: FAS; (n)=number of participants with non-missing baseline and respective post-baseline value (Week 1, Week 4 [LOCF], or Week 12 [LOCF]) for placebo, tolterodine ER, and fesoterodine, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 448 | 926 | 908
percentage of participants
  Week 1 (n=422, 911, 899) | 17.6 | 24.5 | 25.1
  Week 4 [LOCF] (n=448, 922, 908) | 39.5 | 46.7 | 51.1
  Week 12 [LOCF] (n=448, 926, 908) | 53.8 | 58.1 | 63.2
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment difference in continent rate for fesoterodine vs placebo at Week 1; Test type: Superiority or Other; p = 0.0008, Cochran-Mantel-Haenszel; P-value based on Cochran-Mantel-Haenszel test stratified by baseline UUI quartile
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment difference in continent rate for Tolterodine ER vs placebo at Week 1; Test type: Superiority or Other; p = 0.0024, Cochran-Mantel-Haenszel; P-value based on Cochran-Mantel-Haenszel test stratified by baseline UUI quartile
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference in continent rate for fesoterodine vs Tolterodine ER at Week 1; Test type: Superiority or Other; p = 0.6514, Cochran-Mantel-Haenszel; P-value based on Cochran-Mantel-Haenszel test stratified by baseline UUI quartile
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Treatment difference in continent rate for fesoterodine vs placebo at Week 4; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; P-value based on Cochran-Mantel-Haenszel test stratified by baseline UUI quartile
Statistical Analysis 5: Comparison: Placebo vs Tolterodine ER; Treatment difference in continent rate for Tolterodine ER vs placebo at Week 4; Test type: Superiority or Other; p = 0.0063, Cochran-Mantel-Haenszel; P-value based on Cochran-Mantel-Haenszel test stratified by baseline UUI quartile
Statistical Analysis 6: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference in continent rate for fesoterodine vs Tolterodine ER at Week 4; Test type: Superiority or Other; p = 0.0494, Cochran-Mantel-Haenszel; P-value based on Cochran-Mantel-Haenszel test stratified by baseline UUI quartile
Statistical Analysis 7: Comparison: Placebo vs Fesoterodine; Treatment difference in continent rate for fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p = 0.0003, Cochran-Mantel-Haenszel; P-value based on Cochran-Mantel-Haenszel test stratified by baseline UUI quartile
Statistical Analysis 8: Comparison: Placebo vs Tolterodine ER; Treatment difference in continent rate for Tolterodine ER vs placebo at Week 12; Test type: Superiority or Other; p = 0.0991, Cochran-Mantel-Haenszel; P-value based on Cochran-Mantel-Haenszel test stratified by baseline UUI quartile
Statistical Analysis 9: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference in continent rate for fesoterodine vs Tolterodine ER at Week 12; Test type: Superiority or Other; p = 0.0169, Cochran-Mantel-Haenszel; P-value based on Cochran-Mantel-Haenszel test stratified by baseline UUI quartile

16. Secondary Outcome: Change From Baseline in Patient Perception of Bladder Condition (PPBC)
Description: Number of participants in 4-point category: ≥2 points improvement (major improvement; negative change from baseline); 1 point improvement (minor improvement); no change; deterioration (positive change from baseline), based on PPBC score (rated on 6-point scale: 1=no problems at all; 6=many severe problems). Score change: score at observation minus score at baseline; re-scaled to 4-point categorical variables.
Time Frame: Baseline, Week 1, Week, 4, Week 12
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 455 | 937 | 918
participants
  Week 1 (n=452, 931, 913) ≥2 points improvement | 43 | 138 | 144
  Week 1: 1-point improvement | 144 | 278 | 280
  Week 1: no change | 210 | 434 | 428
  Week 1: deterioration | 55 | 81 | 61
  Week 4 (n=455, 937, 918) ≥2 points improvement | 111 | 290 | 334
  Week 4: 1-point improvement | 124 | 298 | 280
  Week 4: no change | 172 | 285 | 250
  Week 4: deterioration | 48 | 64 | 54
  Week 12 (n=455, 937, 918) ≥2 points improvement | 166 | 379 | 440
  Week 12: 1-point improvement | 106 | 250 | 236
  Week 12: no change | 133 | 249 | 189
  Week 12: deterioration | 50 | 59 | 53
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 1; Test type: Superiority or Other; p = 0.0009, Cochran-Mantel-Haenszel; P-value was obtained from a Cochran-Mantel-Haenszel test (CMH) with modified ridit scoring and stratified by country
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 1; Test type: Superiority or Other; p = 0.0279, Cochran-Mantel-Haenszel; P-value was obtained from a Cochran-Mantel-Haenszel test (CMH) with modified ridit scoring and stratified by country
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference Tolterodine ER vs Fesoterodine at Week 1; Test type: Superiority or Other; p = 0.2817, Cochran-Mantel-Haenszel; P-value was obtained from a Cochran-Mantel-Haenszel test (CMH) with modified ridit scoring and stratified by country
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 4; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; P-value was obtained from a Cochran-Mantel-Haenszel test (CMH) with modified ridit scoring and stratified by country
Statistical Analysis 5: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 4; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; P-value was obtained from a Cochran-Mantel-Haenszel test (CMH) with modified ridit scoring and stratified by country
Statistical Analysis 6: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference Tolterodine ER vs Fesoterodine at Week 4; Test type: Superiority or Other; p = 0.0177, Cochran-Mantel-Haenszel; P-value was obtained from a Cochran-Mantel-Haenszel test (CMH) with modified ridit scoring and stratified by country
Statistical Analysis 7: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; P-value was obtained from a Cochran-Mantel-Haenszel test (CMH) with modified ridit scoring and stratified by country
Statistical Analysis 8: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 12; Test type: Superiority or Other; p = 0.0107, Cochran-Mantel-Haenszel; P-value was obtained from a Cochran-Mantel-Haenszel test (CMH) with modified ridit scoring and stratified by country
Statistical Analysis 9: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference Tolterodine ER vs Fesoterodine at Week 12; Test type: Superiority or Other; p = 0.0005, Cochran-Mantel-Haenszel; P-value was obtained from a Cochran-Mantel-Haenszel test (CMH) with modified ridit scoring and stratified by country

17. Secondary Outcome: Change From Baseline in Urgency Perception Scale (UPS). UPS Formerly Known as Patient Perception of Urgency Scale (PPUS) in the Protocol.
Description: Number of participants in 3-point category: improvement [≥1-point improvement]; no change; deterioration [≥1-point decrease], based on UPS score (rated on 3-point scale: 1=not able to hold urine; 3=able to finish what I am doing). Score change calculated as score at observation minus score at baseline; re-scaled to 3-point categorical variables.
Time Frame: Baseline, Week 1, Week, 4, Week 12
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 455 | 938 | 918
participants
  Week 1 (n=452, 932, 913) improvement | 97 | 264 | 267
  Week 1: no change | 326 | 619 | 609
  Week 1: deterioration | 29 | 49 | 37
  Week 4 (n=455, 938, 918) improvement | 161 | 376 | 421
  Week 4: no change | 271 | 511 | 467
  Week 4: deterioration | 23 | 51 | 30
  Week 12 (n=455, 938, 918) improvement | 183 | 440 | 495
  Week 12: no change | 239 | 455 | 393
  Week 12: deterioration | 33 | 43 | 30
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 1; Test type: Superiority or Other; p = 0.0011, Cochran-Mantel-Haenszel; P-value was obtained from a Cochran-Mantel-Haenszel test (CMH) with modified ridit scoring and stratified by country
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 1; Test type: Superiority or Other; p = 0.0072, Cochran-Mantel-Haenszel; P-value was obtained from a Cochran-Mantel-Haenszel test (CMH) with modified ridit scoring and stratified by country
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference fesoterodine vs Tolterodine ER at Week 1; Test type: Superiority or Other; p = 0.3713, Cochran-Mantel-Haenszel; P-value was obtained from a Cochran-Mantel-Haenszel test (CMH) with modified ridit scoring and stratified by country
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 4; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel; P-value was obtained from a Cochran-Mantel-Haenszel test (CMH) with modified ridit scoring and stratified by country
Statistical Analysis 5: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 4; Test type: Superiority or Other; p = 0.1485, Cochran-Mantel-Haenszel; P-value was obtained from a Cochran-Mantel-Haenszel test (CMH) with modified ridit scoring and stratified by country
Statistical Analysis 6: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference fesoterodine vs Tolterodine ER at Week 4; Test type: Superiority or Other; p = 0.0040, Cochran-Mantel-Haenszel; P-value was obtained from a Cochran-Mantel-Haenszel test (CMH) with modified ridit scoring and stratified by country
Statistical Analysis 7: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; P-value was obtained from a Cochran-Mantel-Haenszel test (CMH) with modified ridit scoring and stratified by country
Statistical Analysis 8: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 12; Test type: Superiority or Other; p = 0.0060, Cochran-Mantel-Haenszel; P-value was obtained from a Cochran-Mantel-Haenszel test (CMH) with modified ridit scoring and stratified by country
Statistical Analysis 9: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference fesoterodine vs Tolterodine ER at Week 12; Test type: Superiority or Other; p = 0.0016, Cochran-Mantel-Haenszel; P-value was obtained from a Cochran-Mantel-Haenszel test (CMH) with modified ridit scoring and stratified by country

18. Secondary Outcome: Change From Baseline in Overactive Bladder Questionnaire (OAB-q): Symptom Bother Score at Week 12
Description: Symptom bother score derived as sum of scores for questions 1-8; lowest possible raw score: 8; highest possible score: 48. Data analyzed based on transformation of the score to a 0 to 100 scale [(Actual total raw score - lowest possible value of raw score)/range]*100. Higher scores values indicative of greater symptom bother. Negative change in Symptom Bother Score indicates improvement.
Time Frame: Baseline, Week 12
Population: FAS; (n)=number of participants with non-missing numerical change from baseline to the respective post-baseline value (Week 12 [LOCF]) for placebo, tolterodine ER, and fesoterodine, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 436 | 897 | 876
scores on a scale | -21.8 (1.3) | -24.3 (1.0) | -28.9 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment difference fesoterodine vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -7.1, 95% CI 2-sided [-9.5 to -4.7], Standard Error of Mean 1.2 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment difference Tolterodine ER vs placebo at Week 12; Test type: Superiority or Other; p = 0.0458, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-4.8 to -0.0], Standard Error of Mean 1.2 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment difference Tolterodine ER vs Fesoterodine at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = -4.6, 95% CI 2-sided [-6.6 to -2.7], Standard Error of Mean 1.0 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean

19. Secondary Outcome: Change From Baseline in Overactive Bladder Questionnaire (OAB-q): Health Related Quality of Life (HRQL) at Week 12
Description: HRQL domain and total raw score derived as sum of scores (6-point scale:
  1=not at all/none of the time; 6=a very great deal/all of the time). Transformed score (Total HRQL or domain)=[(Highest possible raw score- Actual total raw score)/Raw score range] * 100. Higher transformed scores indicative of better HRQL. Positive change in HRQL Score indicates improvement.
Time Frame: Baseline, Week 12
Population: as for outcome 18
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 435 | 894 | 875
scores on a scale
  HRQL scale score total (n=431, 892, 873) | 17.2 (1.2) | 19.5 (1.0) | 22.9 (1.0)
  HRQL concern domain (n=434, 894, 875) | 20.2 (1.4) | 22.5 (1.1) | 26.8 (1.1)
  HRQL coping domain (n=433, 892, 875) | 19.0 (1.4) | 22.0 (1.1) | 25.9 (1.2)
  HRQL sleep domain (n=433, 894, 875) | 16.6 (1.3) | 18.7 (1.1) | 21.0 (1.1)
  HRQL social interaction domain (n=435, 894, 873) | 10.8 (1.0) | 12.0 (0.8) | 13.9 (0.8)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo: HRQL scale score total; Test type: Superiority or Other; p < 0.0001, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = 5.6, 95% CI 2-sided [3.4 to 7.9], Standard Error of Mean 1.1 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs Placebo: HRQL scale score total; Test type: Superiority or Other; p = 0.0429, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = 2.3, 95% CI 2-sided [0.1 to 4.6], Standard Error of Mean 1.1 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 3: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER: HRQL scale score total; Test type: Superiority or Other; p = 0.0003, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = 3.3, 95% CI 2-sided [1.5 to 5.2], Standard Error of Mean 0.9 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo: HRQL concern domain; Test type: Superiority or Other; p < 0.0001, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = 6.6, 95% CI 2-sided [4.0 to 9.2], Standard Error of Mean 1.3
Statistical Analysis 5: Comparison: Placebo vs Tolterodine ER; Treatment Difference Placebo vs Tolterodine ER: HRQL concern domain; Test type: Superiority or Other; p = 0.0795, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = 2.3, 95% CI 2-sided [-0.3 to 4.9], Standard Error of Mean 1.3 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 6: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER: HRQL concern domain; Test type: Superiority or Other; p < 0.0001, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = 4.2, 95% CI 2-sided [2.1 to 6.3], Standard Error of Mean 1.1 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 7: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo: HRQL coping domain; Test type: Superiority or Other; p < 0.0001, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = 7.0, 95% CI 2-sided [4.3 to 9.6], Standard Error of Mean 1.4 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 8: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo: HRQL coping domain; Test type: Superiority or Other; p = 0.0229, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = 3.1, 95% CI 2-sided [0.4 to 5.7], Standard Error of Mean 1.3 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 9: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Fesoterodine vs Tolterodine ER: HRQL coping domain; Test type: Superiority or Other; p = 0.0004, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = 3.9, 95% CI 2-sided [1.7 to 6.0], Standard Error of Mean 1.1 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 10: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo: HRQL sleep domain; Test type: Superiority or Other; p = 0.0003, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = 4.5, 95% CI 2-sided [2.0 to 6.9], Standard Error of Mean 1.2 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 11: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo: HRQL sleep domain; Test type: Superiority or Other; p = 0.0923, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [-0.3 to 4.5], Standard Error of Mean 1.2 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 12: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Tolterodine ER vs Fesoterodine: HRQL sleep domain; Test type: Superiority or Other; p = 0.0180, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [0.4 to 4.4], Standard Error of Mean 1.0 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 13: Comparison: Placebo vs Fesoterodine; Treatment Difference Fesoterodine vs placebo: HRQL social interaction domain; Test type: Superiority or Other; p = 0.0011, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = 3.2, 95% CI 2-sided [1.3 to 5.1], Standard Error of Mean 1.0 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 14: Comparison: Placebo vs Tolterodine ER; Treatment Difference Tolterodine ER vs placebo: HRQL social interaction domain; Test type: Superiority or Other; p = 0.2208, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-0.7 to 3.1], Standard Error of Mean 1.0 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean
Statistical Analysis 15: Comparison: Tolterodine ER vs Fesoterodine; Treatment Difference Tolterodine ER vs Fesoterodine: HRQL social interaction domain; Test type: Superiority or Other; p = 0.0117, ANCOVA; Based on an analysis of covariance model with terms for country and treatment and with baseline value as a covariate; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [0.4 to 3.5], Standard Error of Mean 0.8 — Treatment difference LSMean difference (SE), SE is recorded as parameter dispersion type: standard error of the mean

20. Post Hoc Outcome: Post-hoc Adverse Events (AEs)
Description: An adverse event is any untoward medical occurrence in a clinical investigation in which the participant was administered a product or medical device; the event does not necessarily need to have a causal relationship with the treatment or usage.
Time Frame: Baseline up to Week 12
Population: Safety population included all participants who were randomized and received at least 1 dose of study treatment. N=number of participants with AEs noted in other unreviewed medical chart records as performed at other departments during the clinical trial but were not included as AEs in Case Report Forms; reported post-hoc.
Measure: Number; unit: events
Arm/Group | Tolterodine ER | Fesoterodine
Number analyzed (Participants) | 1 | 1
events
  Constipation | 1 | 0
  Fingers tingling | 0 | 1
  Finger numbness | 0 | 1
  Hypertension | 0 | 2
  Diabetes mellitus | 0 | 2
  Abdominal distension and discomfort | 0 | 1
  Tina pedis | 0 | 1
  Tingling sensation/decreased sensation of fingers | 0 | 1
  Dyspepsia | 0 | 1
  Abdominal bloating | 0 | 1

ADVERSE EVENTS:
Description: An Adverse Event (AE) term may be reported as both a serious and non-serious AE, but are distinct events. AE may = serious for 1 subject and = non-serious for another subject or subject may have experienced both a serious and non-serious episode of the same event.
Arm/Group | Placebo | Tolterodine ER | Fesoterodine
Serious Adverse Events (participants affected / at risk) | 8/478 | 6/973 | 13/960
Other Adverse Events (participants affected / at risk) | 83/478 | 261/973 | 375/960
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=478) | Tolterodine ER (N=973) | Fesoterodine (N=960)
Angina unstable (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Mitral valve stenosis (Cardiac disorders) | 1 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 1
Mania (Psychiatric disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Allergic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Cholecystectomy (Surgical and medical procedures) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=478) | Tolterodine ER (N=973) | Fesoterodine (N=960)
Constipation (Gastrointestinal disorders) | 7 | 30 | 42
Diarrhoea (Gastrointestinal disorders) | 3 | 11 | 11
Dry mouth (Gastrointestinal disorders) | 26 | 130 | 265
Dyspepsia (Gastrointestinal disorders) | 2 | 10 | 21
Nausea (Gastrointestinal disorders) | 3 | 13 | 11
Oedema peripheral (General disorders) | 5 | 14 | 4
Bronchitis (Infections and infestations) | 6 | 10 | 3
Influenza (Infections and infestations) | 1 | 12 | 5
Nasopharyngitis (Infections and infestations) | 6 | 9 | 8
Sinusitis (Infections and infestations) | 2 | 11 | 4
Urinary tract infection (Infections and infestations) | 5 | 12 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 9 | 8
Headache (Nervous system disorders) | 6 | 20 | 27
Dysuria (Renal and urinary disorders) | 2 | 8 | 10
Polyuria (Renal and urinary disorders) | 10 | 24 | 29
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 12
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.